CLINICAL TRIAL: NCT02253745
Title: A Double-blind, Randomized, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Repeat Oral Doses of V81444 in Volunteers With Attention Deficit / Hyperactivity Disorder (ADHD)
Brief Title: Safety, Tolerability, PK & Efficacy of V81444 in Volunteers With Attention Deficit/ Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V81444-1CNS-01
Record Dates: First submitted 2014-09-26; First posted 2014-10-01 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2015-12

CONDITIONS: ADHD
Keywords: ADHD; Attention Deficit/ Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo:V81444 (Experimental): Placebo followed by a 7 day washout then V81444
  Interventions: Drug: V81444; Drug: Placebo
- V81444:placebo (Experimental): V81444 followed by a 7 day washout then Placebo
  Interventions: Drug: V81444; Drug: Placebo

INTERVENTIONS:
Drug: V81444 — V81444 capsules for oral administration, 100 mg twice daily for 13 days and once on Day 14
Drug: Placebo — Capsules to match V81444 twice daily for 13 days and once on Day 14

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability, effectiveness, and pharmacokinetics (PK) of twice daily oral doses of V81444 in adults with ADHD. Pharmacokinetics (PK) is the study of how a drug is absorbed, distributed, metabolized, and eventually eliminated by the body. Pharmacokinetics is what the body does to the drug. Blood samples will be taken throughout the study for PK analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  1. Be male or female subjects aged 18 to 50 years inclusive
  2. Meet DSM-IV-TR criteria for a primary diagnosis of ADHD combined, hyperactive-impulsive or predominantly inattentive type; confirmed by a minimum score of 24 on the ADHD-RS with adult prompts:
  3. Have a body mass index (BMI) between 19 and 32 kg/m2 inclusive
  4. Be willing and able to comply with the requirements of the entire study
  5. Be able to read and understand English
  6. Give written informed consent

Exclusion Criteria:

1. Have a significant medical condition or a history of such a condition that the Investigator considers should exclude the subject from the study
2. Have any other significant psychiatric disorder, as determined by the Structured Clinical Interview for DSM-IV-TR Axis I Disorders (SCID-I)
3. Have known mental impairment defined as an intelligence quotient (IQ) less than 75, or clinical evidence of mental impairment based on the opinion of the Investigator
4. Have a history or evidence of clinically significant GI disease, including ulcers, gastro-esophageal reflux disease, hiatus hernia or gastritis
5. Have had any previous gastric surgery and/or bariatric procedure
6. Have any known malformations that would make EGD difficult or unsafe
7. Have taken any prohibited concomitant medication
8. Have multiple drug allergies or be allergic to any of the components of V81444 study medication or its matching placebo (see Section 7.1) or lidocaine
9. Have abused drugs in the 12 months before study drug administration
10. In the 90 days before study drug administration, on average

    * have smoked more than 5 cigarettes per day
    * have consumed more than 28 units of alcohol per week
    * have consumed more than 500 mg of caffeine per day
11. In the 2 calendar months before study drug administration

    * have donated blood or plasma in excess of 500 mL
    * been exposed to any new investigational agent
12. In the calendar month prior to screening

    * used non-steroidal anti-inflammatory drugs regularly
    * had a new tattoo or body piercing
13. Have any clinically relevant abnormal findings at Screening and/or admission
14. Plan to undergo elective procedures/surgery at any time during the study
15. Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
ADHD-RS | 5 weeks
  The absolute and change from baseline in ADHD-RS scores, and percentage change from baseline in ADHD-RS score will be summarized appropriately

SECONDARY OUTCOMES:
PERM-P | 5 weeks
  The average of the on-treatment total post-dose PERM-P scores for each treatment assessment day during the randomized treatment period will be calculated for each individual.
Clinical Global Impression (CGI) | 5 weeks
  The CGI scores will be summarised using frequency counts and percentages.
Safety and Tolerability | 11 weeks
  Parameters for evaluation of safety and tolerability:
  Adverse events, Clinical laboratory safety tests, Physical examination, Vital signs, 12-lead ECG, Telemetry, EGD findings, CSSRS, LSEQ

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Vince, MD, Principal Investigator — VACR
Locations (1):
- Vince and Associates Clinical Research, Kansas City, Kansas, United States